CLINICAL TRIAL: NCT02583854
Title: Comparison Study of Compression Devices Used in Transradial Coronary Angiography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Helse Sor-Ost (Other Government)
Responsible Party: Principal Investigator, Anders Opdahl, MD, PhD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 573099
Record Dates: First submitted 2015-10-21; First posted 2015-10-22 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Peripheral Artery Occlusion; Hemostasis; Injury of Radial Artery
Keywords: Coronary angiography; Transradial; Patient experience; VAS; Compression device

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hemostasis achieved by TR Band (Active Comparator): After the transradial procedure and randomization TR Band will be applied to achieve hemostasis. Patient experience and complications after the application will be measured.
  Interventions: Device: TR-Band, Terumo
- Hemostasis achieved by RY Stop (Experimental): After the transradial procedure and randomization, RY Stop will be applied to achieve hemostasis. Patient experience and complications after the application will be measured.
  Interventions: Device: RY-STOP hemostasis device

INTERVENTIONS:
Device: RY-STOP hemostasis device
  Arms: Hemostasis achieved by RY Stop
Device: TR-Band, Terumo
  Arms: Hemostasis achieved by TR Band

SUMMARY:
The transradial route is used in 90% of the coronary angiograms performed at Oslo University Hospital (OUS), Ullevål. A compression device needs to be applied after the procedure to achieve hemostasis. Patients and staff will benefit from using a device that yields safe and painless hemostasis.

Patients will be randomly assigned to receive either the standard compression device (control group, A) or a recently developed compression device (experimental group, B). The study will be designed as a non-inferiority, prospective randomized controlled trial, with outcome measures being patient comfort during compression time and complication rates. Complications that will be measured are radial artery occlusion (RAO) measured using ultrasound at a follow up visit. Hematomas or bleeds from the puncture site after application of the compression device will also be classified as complications.

The aim of the study is to investigate whether the new device, RY-STOP is non-inferior compared to the standard device, when considering the outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing coronary angiograms via the transradial route

Exclusion Criteria:

* Patients who have a long way to travel for the follow up, ultrasound scan
* Patients that do not understand Norwegian
* Patients presenting with acute ST segment elevation myocardial infarction (STEMI)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 499 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Radial artery occlusion | 90-120 days
  Subjects wil have an ultrasound scan of their radial artery preformed after their transradial coronary angiogram to see the rate of occluded arteries.

SECONDARY OUTCOMES:
Patient experience | 1-4 hours
  Patients will be asked to rate their comfort level associated with the hemostasis device they have been assigned
Device complications | 1-4 hours
  Staff responsible for the application of the hemostasis devices will be asked to observe and record bleeds and hematomas that occur.

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Due-Tonnessen N, Egeland CH, Meyerdierks OJ, Opdahl A. Is radial artery occlusion and local vascular complications following transradial coronary procedures affected by the type of haemostasis device used? A non-inferiority Randomized Controlled Trial (RadCom trial). Eur J Cardiovasc Nurs. 2021 Aug 20;20(6):580-587. doi: 10.1093/eurjcn/zvab004. PMID 33615328